CLINICAL TRIAL: NCT06133686
Title: Implementing Oral (Event-driven and Daily) and Long-acting Pre-Exposure Prophylaxis in Mobile Men in Sub-Saharan Africa: a Phase 3b, Open-label, Hybrid Type 2 Implementation and Effectiveness Trial
Brief Title: Implementing Oral (Event-driven and Daily) and Long-acting Pre-Exposure Prophylaxis in Mobile Men in Sub-Saharan Africa
Acronym: MOBILEMEN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: King's College London (Other); London School of Hygiene and Tropical Medicine (Other); Africa Health Research Institute (Other); Wits Health Consortium (Pty) Ltd (Other); University College, London (Other); Ministry of Health, Uganda (Other Government); Desmond Tutu HIV Foundation (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RGDER231010
Record Dates: First submitted 2023-10-19; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: HIV
Keywords: Mobile Men; HIV; Pre-exposure prophylaxis; Truvada; Cabotegravir
MeSH Terms: interventions — Tenofovir; Emtricitabine; cabotegravir

STUDY DESIGN:
Intervention Model Description: This is a Phase 3b, open label, hybrid type 2 study with co-primary aims of effective use and implementation. This is a mixed method, multi-setting, multi-country randomized controlled trial, carried out in South Africa and Uganda to compare persistence in care for oral PrEP and CAB-LA in mobile men, which will inform PrEP implementation in men. Mobile men aged 18+ years, will be recruited from outreach settings in in South Africa and Uganda. Those testing HIV negative (target sample size, n=400) will be randomized into 2 groups: Group A will receive oral TDF-FTC PrEP (using either event-driven or daily) and Group B will receive CAB-LA over 9-months. After 9- months participants from both groups will be offered choice of PrEP for a further 9-months, with the ability to change choice as required. Switch PrEP options will be monitored. Those receiving oral PrEP will be able to choose between event-driven and daily PrEP with the emphasis on coital coverage by PrEP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Other): Oral Tenofovir disoproxil fumarate/emtricitabine (TDF-FTC) followed by choice of TDF-FTC or CAB-LA
  Interventions: Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF-FTC), cabotegravir (CAB-LA)
- Group B (Other): Long-acting injectable cabotegravir (CAB-LA) followed by choice of TDF-FTC or CAB-LA
  Interventions: Drug: Cabotegravir (CAB-LA), Tenofovir disoproxil fumarate/emtricitabine (TDF-FTC)

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF-FTC), cabotegravir (CAB-LA) — Group A will receive oral TDF-FTC PrEP (using either event-driven or daily) for 9-months. After 9-months, participants will be offered choice of PrEP (either TDF-FTC or CAB-LA) for a further 9-months, with the ability to change choice as required. Those receiving oral PrEP will be able to choose between event-driven and daily PrEP with the emphasis on coital coverage by PrEP
  Arms: Group A
Drug: Cabotegravir (CAB-LA), Tenofovir disoproxil fumarate/emtricitabine (TDF-FTC) — Group B will receive CAB-LA for 9-months. After 9-months participants will be offered choice of PrEP (either TDF-FTC or CAB-LA) for a further 9-months, with the ability to change choice as required. Those receiving oral PrEP will be able to choose between event-driven and daily PrEP with the emphasis on coital coverage by PrEP.
  Arms: Group B

SUMMARY:
Title: Implementing oral (event-driven and daily) and long-acting Pre-exposure prophylaxis (PrEP) in mobile men in Sub-Saharan Africa

Design: A mixed method, multi-setting, multi-country, phase 3b, open-label, hybrid type 2 implementation and effectiveness randomized controlled trial (RCT). The trial will be carried out in 400 HIV negative men aged 18+ years in South Africa and Uganda. Men will be randomized 1:1 to either Group A: oral Tenofovir disoproxil fumarate/emtricitabine (TDF-FTC) PrEP (event-driven or daily) or Group B: Long-acting injectable cabotegravir (CAB-LA) over 9-months. After 9-months participants from both groups will be offered choice of PrEP (oral TDF-FTC or CAB-LA) for a further 9-months, with the ability to change choice as required. Various strategies to support PrEP adoption, initiation, and persistence will be implemented, monitored, and reported on using a RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) implementation science framework.

Treatment: CAB-LA or oral TDF-FTC Duration: 18 months

DETAILED DESCRIPTION:
BACKGROUND HIV prevention pre-exposure prophylaxis (PrEP) has not been evaluated in men who mainly have sex with women and who may be at high risk of HIV acquisition due to high HIV prevalence in partners or particularly risky behaviours. Research to fill these data gaps is required to facilitate their inclusion in PrEP guidelines. Furthermore, with increasing PrEP options, recommendations to users and providers in high-burden / resource constrained settings is a key focus of the Sustainable Development Goal target to end AIDS by 2030. To date, HIV prevention research has largely focussed on adolescent girls and young women (AGYW) in low and middle income countries and men who have sex with men (MSM) in high income countries. Research on the user experience and choice of oral PrEP or CAB-LA PrEP amongst vulnerable heterosexual men is required.

Men consistently fare worse than women in levels of HIV testing and ART initiation with significant challenges in sub-Saharan Africa (SSA) for engagement and persistence in HIV treatment programmes well described. Despite this, heterosexual men represent the largest unaddressed gap in HIV services in SSA. Indeed, the failure of Treatment As Prevention trials (TASP) to show effect was in the main due to the failure to test and treat young men. Men who are mobile for work or through looking for work, are viewed by the WHO as a key population at high risk for HIV. As Africa's large youth bulge moves into young adulthood, the search for work and consequent mobile lifestyles will further increase.

In order to improve uptake, persistence, and effective use of all forms of PrEP, there is a need for simplified and differentiated delivery of PrEP that is person- and community-centred specifically for men. Effective use requires that all sex acts are covered by an effective prevention intervention such as PrEP. Given the importance of flexibility due to travel in this group, our hypothesis is that both oral PrEP (in particular, event-driven) and CAB-LA PrEP will be highly acceptable to men in two high-burden, resource limited, African countries, with high levels of effective use including persistence and coital coverage.

This is the first multi-country PrEP study for implementing both event-driven oral PrEP and Long-acting injectable cabotegravir (CAB-LA) in men in SSA (South Africa and Uganda). The programme will provide the evidence and cost-effectiveness analysis which is critical to decision making by African governments and donors on how to prioritise prevention resources and inform guidelines.

STUDY OBJECTIVES Effective use is defined as PrEP uptake and persistence, retention in care, and HIV exposure coverage with adequate drug tissue levels.

Overall Objective To assess effectiveness and implementation of CAB-LA and oral TDF-FTC (both daily and event driven) through comparison of uptake, retention in care, coital coverage, and participant choice

Primary Objective

1. Primary user effectiveness objective: To compare short term (9 months) and longer term (18 months) PrEP persistence patterns across different PrEP modalities (oral and injectable) amongst men who are mobile for work in South Africa and Uganda.
2. Primary implementation objective: To compare adoption (uptake and choice) across the different PrEP modalities (oral and injectable) amongst men who are mobile for work in South Africa and Uganda.

Adoption is defined as 1) uptake: do people accept and use the intervention they're randomised to, and 2) choice: based on the post-randomised period, i.e., months 9-18, what PrEP do they choose)

Secondary clinical objectives

1. To compare the effective coital coverage of oral daily/on-demand oral TDF-FTC versus CAB-LA
2. To describe the safety, tolerability and acceptance of all methods, as determined by self-reported adverse side effects, AEs and reasons for PrEP pause or discontinuation.

Secondary implementation objectives:

1. To understand the Reach of PrEP for mobile men and understand the barriers to and facilitators of uptake amongst those at risk who do and do not accept oral or LA PrEP.
2. To describe adoption:

   1. To identify characteristics of men who adopt oral PrEP versus CAB-LA
   2. To describe patterns of use of daily, on-demand, and long-acting PrEP amongst different groups of mobile men.
3. To understand the implementation of on-demand and long-acting PrEP for mobile men amongst service providers to inform scale-up.

   1. To understand the feasibility and fidelity of delivering on-demand and long-acting PrEP in different settings.
   2. To describe how on-demand and long-acting PrEP are delivered in practice.
   3. To describe the service-level needs to implement on-demand and long-acting PrEP.
   4. To evaluate acceptabiltiy and implementation of antibody based monitoring HIV status for CAB-LA.
4. To assess the total and average cost of oral PrEP and CAB-LA in South Africa and Uganda under study conditions from the provider perspective (Maintenance).

Exploratory objectives

1. To describe HIV incidence across the two PrEP modality arms
2. To describe any evidence of HIV drug resistance mutations in participants who acquire HIV infection whilst using PrEP across the two PrEP modality arms.
3. To describe persistence in care of those diagnosed HIV infected at screening.
4. To describe body mass index (BMI) and blood pressure across both arms.

STUDY DESIGN We will use a hybrid effectiveness implementation type 2 trial to evaluate the initial implementation (scale-up) phase of CAB-LA as a PrEP option in men who are mobile for work in South Africa and Uganda with a high burden of HIV. This is a Phase 3b, open label, hybrid type 2 study with co-primary aims of effective use and implementation.

This is a mixed method, multi-setting, multi-country randomized controlled trial (RCT), carried out in South Africa and Uganda to compare persistence in care for oral PrEP and CAB-LA in mobile men, which will inform PrEP implementation in men. Mobile men aged 18+ years, will be recruited from outreach settings in South Africa and Uganda. Those testing HIV negative (target sample size, n=400) will be randomized into 2 groups: Group A will receive oral TDF-FTC PrEP (using either event-driven or daily) and Group B will receive CAB-LA over 9-months. After 9- months participants from both groups will be offered choice of PrEP for a further 9-months, with the ability to change choice as required. Switch PrEP options will be monitored. Those receiving oral PrEP will be able to choose between event-driven and daily PrEP with the emphasis on coital coverage by PrEP.

Implementation Framework: The project utilises the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, and Maintenance) to evaluate MOBILE MEN's PrEP delivery preferences and patterns of use.

Participants will be supported in taking PrEP and the social science and implementation science data collection will feedback findings in real time, on the ways to facilitate men to maximise their adherence to PrEP.

Healthcare providers will be trained to deliver oral (daily and event driven) and injectable PrEP, develop services which are mobile men friendly- non-judgemental, timing and location appropriate for men.

Data will be collected in Uganda and South Africa.

Recruitment settings:

A decentralized model of care for recruitment and persistence in ongoing study will be developed whereby study visits will be conducted through mobile and outreach clinics. Demand creation for PrEP will take place through a community engagement campaign and peer outreach activities prior to the study starting, whereby men in the communities are exposed to PrEP educational materials and encouraged to visit community and public health sites to access sexual health services, including PrEP. Potential participants will be provided with educational information about each of the PrEP products through both the enrolment visit and as part of a community-wide demand creation campaign which precedes the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent
2. Aged 18 years and above on the day of screening
3. Willing to have a HIV test and receive the test results
4. Male at birth
5. In the past 6-months has travelled for work or to find work and spent at least one night away from home for work related purposes.
6. Available for follow up for the duration of the study

Exclusion Criteria:

1. Known HIV infection
2. Confirmed HIV-positive test result, indeterminate HIV test result, and/or signs and symptoms of an acute HIV infection
3. Body weight less than 35Kg at baseline
4. Allergy to any of the study products
5. Medical, social or other condition that, in the opinion of the site investigator, would interfere with the conduct of the study or safety of the participant (e.g., provided by self-report, or found upon medical history and examination or in available medical records)
6. Use of contraindicated medications: Medication for tuberculosis (Rifampin, rifapentine) or anticonvulsants (Carbamazepine, oxcarbazepine, phenobarbital, phenytoin)
7. Other reasons at the discretion of site investigator for unsuitability for study inclusion

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
The primary user effectiveness outcome will be the persistent use of PrEP in the randomised period and throughout the full follow-up period. | 18 months
  Persistence will be a binary outcome capturing whether a participant has used PrEP persistently or not. For participants receiving CAB-LA, this will be based on whether they received all injections as per schedule or not. For participants receiving TDF-FTC, this will be based on whether they have attended scheduled visits, had TDF-FTC dispensed, and have detectable TFV-DP levels in dried blood spots.
The primary implementation outcome will be PrEP adoption | 18 months
  PrEP adoption was assessed as uptake of PrEP in months 0-9. This is a binary variable that will capture whether or not a participant was offered and took up the offer of PrEP during the 9-month randomized period.
The primary implementation outcome will be PrEP adoption | 18 Months
  PrEP adoption was assessed as the choice preference of PrEP in months 9-18. This is a categorical variable that will measure the proportions that choose and uptake each modality (daily or event-driven TDF-FTC or CAB-LA) captured at the start and the end of the subsequent 9-month choice period

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Ruzagira, PhD, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit; Julie Fox, PhD, Study Chair — King's College London

IPD SHARING:
Plan to Share IPD: Yes
The team is committed to open access data. The results of the study and anonymized data sets will be published in open access peer-reviewed journals and data repositories.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Zhang J, Li C, Xu J, Hu Z, Rutstein SE, Tucker JD, Ong JJ, Jiang Y, Geng W, Wright ST, Cohen MS, Shang H, Tang W. Discontinuation, suboptimal adherence, and reinitiation of oral HIV pre-exposure prophylaxis: a global systematic review and meta-analysis. Lancet HIV. 2022 Apr;9(4):e254-e268. doi: 10.1016/S2352-3018(22)00030-3. PMID 35364026
- [Background] Giguere K, Eaton JW, Marsh K, Johnson LF, Johnson CC, Ehui E, Jahn A, Wanyeki I, Mbofana F, Bakiono F, Mahy M, Maheu-Giroux M. Trends in knowledge of HIV status and efficiency of HIV testing services in sub-Saharan Africa, 2000-20: a modelling study using survey and HIV testing programme data. Lancet HIV. 2021 May;8(5):e284-e293. doi: 10.1016/S2352-3018(20)30315-5. Epub 2021 Mar 2. PMID 33667411
- [Background] Iwuji CC, Orne-Gliemann J, Larmarange J, Balestre E, Thiebaut R, Tanser F, Okesola N, Makowa T, Dreyer J, Herbst K, McGrath N, Barnighausen T, Boyer S, De Oliveira T, Rekacewicz C, Bazin B, Newell ML, Pillay D, Dabis F; ANRS 12249 TasP Study Group. Universal test and treat and the HIV epidemic in rural South Africa: a phase 4, open-label, community cluster randomised trial. Lancet HIV. 2018 Mar;5(3):e116-e125. doi: 10.1016/S2352-3018(17)30205-9. Epub 2017 Nov 30. PMID 29199100
- [Background] The Global Men and HIV Technical Working Group (MENHT). HIV gap in men. HIV gap in men: the Global Men and HIV Technical Working Group (MENHT) Webinar Series - Episode #4 (who.int) 2021.
- [Background] Delany-Moretlwe S, Hughes JP, Bock P, Ouma SG, Hunidzarira P, Kalonji D, Kayange N, Makhema J, Mandima P, Mathew C, Spooner E, Mpendo J, Mukwekwerere P, Mgodi N, Ntege PN, Nair G, Nakabiito C, Nuwagaba-Biribonwoha H, Panchia R, Singh N, Siziba B, Farrior J, Rose S, Anderson PL, Eshleman SH, Marzinke MA, Hendrix CW, Beigel-Orme S, Hosek S, Tolley E, Sista N, Adeyeye A, Rooney JF, Rinehart A, Spreen WR, Smith K, Hanscom B, Cohen MS, Hosseinipour MC; HPTN 084 study group. Cabotegravir for the prevention of HIV-1 in women: results from HPTN 084, a phase 3, randomised clinical trial. Lancet. 2022 May 7;399(10337):1779-1789. doi: 10.1016/S0140-6736(22)00538-4. Epub 2022 Apr 1. PMID 35378077
- [Background] Abstracts from the 2022 Conference on Retroviruses and Opportunistic Infections. Top Antivir Med. 2022 Mar;30(1s):3-382. No abstract available. PMID 35298110
- [Background] World Health Organization : Differentiated and simplified pre-exposure prophylaxis for HIV prevention: update to WHO implementation guidance. Technical Brief. Geneva: World Health Organization; 2022. Licence: CC BY.
- [Background] Guidelines on Long-Acting Injectable Cabotegravir for HIV Prevention [Internet]. Geneva: World Health Organization; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK586584/ PMID 36417549
- [Background] Philbin MM, Parish C, Kinnard EN, Reed SE, Kerrigan D, Alcaide ML, Cohen MH, Sosanya O, Sheth AN, Adimora AA, Cocohoba J, Goparaju L, Golub ET, Fischl M, Metsch LR. Interest in Long-Acting Injectable Pre-exposure Prophylaxis (LAI PrEP) Among Women in the Women's Interagency HIV Study (WIHS): A Qualitative Study Across Six Cities in the United States. AIDS Behav. 2021 Mar;25(3):667-678. doi: 10.1007/s10461-020-03023-9. PMID 32910351
- [Background] Sued O, Nardi N, Spadaccini L. Key population perceptions and opinions about long-acting antiretrovirals for prevention and treatment: a scoping review. Curr Opin HIV AIDS. 2022 May 1;17(3):145-161. doi: 10.1097/COH.0000000000000734. Epub 2022 Apr 18. PMID 35439789
- [Background] Johnson L, Dorrington R. Thembisa version 4.6: National and Provincial Model Outputs. Thembisa. 2023. Available from: https://www.thembisa.org/content/downloadPage/ProvOutput4_6 (Accessed July 4, 2023).
- [Background] Johnson LF, Dorrington RE, Moolla H. Progress towards the 2020 targets for HIV diagnosis and antiretroviral treatment in South Africa. South Afr J HIV Med. 2017 Jul 27;18(1):694. doi: 10.4102/sajhivmed.v18i1.694. eCollection 2017. PMID 29568630
- [Background] Simbayi L, Zuma K, Zungu N, Moyo S, Marinda E, Jooste S, Mabaso M, Ramlangan S, North A, van Zyl J, Mohlabane N, Dietrich C, Naidoo I, SABSSM V Team. South African national HIV prevalence, incidence, behaviour and communication survey, 2017: towards achieving the UNAIDS 90-90-90 targets [Internet]. 2019 [cited 2021 Apr 4]. Available from: http://repository.hsrc.ac.za/handle/20.500.11910/15052
- [Background] Nglazi MD, van Schaik N, Kranzer K, Lawn SD, Wood R, Bekker LG. An incentivized HIV counseling and testing program targeting hard-to-reach unemployed men in Cape Town, South Africa. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):e28-34. doi: 10.1097/QAI.0b013e31824445f0. PMID 22173039
- [Background] Bazzi AR, Valasek CJ, Streuli SA, Vera CF, Harvey-Vera A, Philbin MM, Biello KB, Roth AM, Strathdee SA, Pines HA. Long-Acting Injectable Human Immunodeficiency Virus Pre-Exposure Prophylaxis Preferred Over Other Modalities Among People Who Inject Drugs: Findings from a Qualitative Study in California. AIDS Patient Care STDS. 2022 Jul;36(7):254-262. doi: 10.1089/apc.2022.0068. Epub 2022 Jun 21. PMID 35727647
- [Background] Gill K, Johnson L, Dietrich J, Myer L, Marcus R, Wallace M, Pidwell T, Mendel E, Fynn L, Jones K, Wiesner L, Slack C, Strode A, Spiegel H, Hosek S, Rooney J, Gray G, Bekker LG. Acceptability, safety, and patterns of use of oral tenofovir disoproxil fumarate and emtricitabine for HIV pre-exposure prophylaxis in South African adolescents: an open-label single-arm phase 2 trial. Lancet Child Adolesc Health. 2020 Dec;4(12):875-883. doi: 10.1016/S2352-4642(20)30248-0. Epub 2020 Oct 24. PMID 33222803
- [Background] Kaewpoowat Q, Chariyalertsak S, Phanuphak N, Ramautarsing RA. Long-acting preexposure prophylaxis in low- and middle-income countries: key considerations for implementation. Curr Opin HIV AIDS. 2022 May 1;17(3):135-144. doi: 10.1097/COH.0000000000000729. Epub 2022 Mar 4. PMID 35439788
- [Background] Pike C, Bekker LG. Interrogating the promise of long-acting HIV pre-exposure prophylaxis. Trends Mol Med. 2023 Feb;29(2):93-98. doi: 10.1016/j.molmed.2022.11.003. Epub 2022 Nov 23. PMID 36435632
- [Background] Global Data Lab. Subnational Human Development Index - South Africa. Global Data Lab. Available from: https://globaldatalab.org/shdi/shdi/ZAF/ (Accessed July 1, 2023).
- [Background] Smits J, Permanyer I. The Subnational Human Development Database. Sci Data. 2019 Mar 12;6:190038. doi: 10.1038/sdata.2019.38. PMID 30860498
- [Background] Suite DH, La Bril R, Primm A, Harrison-Ross P. Beyond misdiagnosis, misunderstanding and mistrust: relevance of the historical perspective in the medical and mental health treatment of people of color. J Natl Med Assoc. 2007 Aug;99(8):879-85. PMID 17722664
- [Background] Cooper SE, Rosenblatt J, Gulick RM. Barriers to Uptake of Long-Acting Antiretroviral Products for Treatment and Prevention of Human Immunodeficiency Virus (HIV) in High-Income Countries. Clin Infect Dis. 2022 Nov 21;75(Suppl 4):S541-S548. doi: 10.1093/cid/ciac716. PMID 36410385
- [Background] McCormack S, Dunn DT, Desai M, Dolling DI, Gafos M, Gilson R, Sullivan AK, Clarke A, Reeves I, Schembri G, Mackie N, Bowman C, Lacey CJ, Apea V, Brady M, Fox J, Taylor S, Antonucci S, Khoo SH, Rooney J, Nardone A, Fisher M, McOwan A, Phillips AN, Johnson AM, Gazzard B, Gill ON. Pre-exposure prophylaxis to prevent the acquisition of HIV-1 infection (PROUD): effectiveness results from the pilot phase of a pragmatic open-label randomised trial. Lancet. 2016 Jan 2;387(10013):53-60. doi: 10.1016/S0140-6736(15)00056-2. Epub 2015 Sep 9. PMID 26364263
- [Background] Molina JM, Capitant C, Spire B, Pialoux G, Cotte L, Charreau I, Tremblay C, Le Gall JM, Cua E, Pasquet A, Raffi F, Pintado C, Chidiac C, Chas J, Charbonneau P, Delaugerre C, Suzan-Monti M, Loze B, Fonsart J, Peytavin G, Cheret A, Timsit J, Girard G, Lorente N, Preau M, Rooney JF, Wainberg MA, Thompson D, Rozenbaum W, Dore V, Marchand L, Simon MC, Etien N, Aboulker JP, Meyer L, Delfraissy JF; ANRS IPERGAY Study Group. On-Demand Preexposure Prophylaxis in Men at High Risk for HIV-1 Infection. N Engl J Med. 2015 Dec 3;373(23):2237-46. doi: 10.1056/NEJMoa1506273. Epub 2015 Dec 1. PMID 26624850
- [Background] Dietrich JJ, Ahmed N, Webb EL, Tshabalala G, Hornschuh S, Mulaudzi M, Atujuna M, Stranix-Chibanda L, Nematadzira T, Ssemata AS, Muhumuza R, Seeley J, Bekker LG, Weiss HA, Martinson N, Fox J; CHAPS team. A multi-country cross-sectional study to assess predictors of daily versus on-demand oral pre-exposure prophylaxis in youth from South Africa, Uganda and Zimbabwe. J Int AIDS Soc. 2022 Aug;25(8):e25975. doi: 10.1002/jia2.25975. PMID 36002910
- [Background] Parikh UM, Mellors JW. How could HIV-1 drug resistance impact preexposure prophylaxis for HIV prevention? Curr Opin HIV AIDS. 2022 Jul 1;17(4):213-221. doi: 10.1097/COH.0000000000000746. PMID 35762376
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Proctor EK, Powell BJ, McMillen JC. Implementation strategies: recommendations for specifying and reporting. Implement Sci. 2013 Dec 1;8:139. doi: 10.1186/1748-5908-8-139. PMID 24289295
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Pilgrim NA, Evans TM, Czarnogorski M. A Layer Plus Approach to Implementation Research and Collaboration for Long-Acting Injectable Preexposure Prophylaxis for HIV Prevention. Health Promot Pract. 2022 Nov;23(6):912-915. doi: 10.1177/15248399211053584. Epub 2022 Jun 17. PMID 35713273
- [Background] King DK, Glasgow RE, Leeman-Castillo B. Reaiming RE-AIM: using the model to plan, implement, and evaluate the effects of environmental change approaches to enhancing population health. Am J Public Health. 2010 Nov;100(11):2076-84. doi: 10.2105/AJPH.2009.190959. Epub 2010 Sep 23. PMID 20864705
- [Background] Mhlongo S, Dietrich J, Otwombe KN, Robertson G, Coates TJ, Gray G. Factors associated with not testing for HIV and consistent condom use among men in Soweto, South Africa. PLoS One. 2013 May 16;8(5):e62637. doi: 10.1371/journal.pone.0062637. Print 2013. PMID 23696786
- [Background] Otwombe K, Dietrich J, Laher F, Hornschuh S, Nkala B, Chimoyi L, Kaida A, Gray GE, Miller CL. Health-seeking behaviours by gender among adolescents in Soweto, South Africa. Glob Health Action. 2015 Feb 2;8:25670. doi: 10.3402/gha.v8.25670. eCollection 2015. PMID 25653113
- [Background] Smith P, Marcus R, Bennie T, Nkala B, Nchabeleng M, Latka MH, Gray G, Wallace M, Bekker LG. What do South African adolescents want in a sexual health service? Evidence from the South African Studies on HIV in Adolescents (SASHA) project. S Afr Med J. 2018 Jul 25;108(8):677-681. doi: 10.7196/SAMJ.2018.v108i8.13013. PMID 30182885
- [Background] Pleuhs B, Quinn KG, Walsh JL, Petroll AE, John SA. Health Care Provider Barriers to HIV Pre-Exposure Prophylaxis in the United States: A Systematic Review. AIDS Patient Care STDS. 2020 Mar;34(3):111-123. doi: 10.1089/apc.2019.0189. Epub 2020 Feb 28. PMID 32109141
- [Background] Pilgrim N, Jani N, Mathur S, Kahabuka C, Saria V, Makyao N, Apicella L, Pulerwitz J. Provider perspectives on PrEP for adolescent girls and young women in Tanzania: The role of provider biases and quality of care. PLoS One. 2018 Apr 27;13(4):e0196280. doi: 10.1371/journal.pone.0196280. eCollection 2018. PMID 29702659
- [Background] Breitenstein SM, Gross D, Garvey CA, Hill C, Fogg L, Resnick B. Implementation fidelity in community-based interventions. Res Nurs Health. 2010 Apr;33(2):164-73. doi: 10.1002/nur.20373. PMID 20198637
- [Background] Birgisson NE, Zhao Q, Secura GM, Madden T, Peipert JF. Preventing Unintended Pregnancy: The Contraceptive CHOICE Project in Review. J Womens Health (Larchmt). 2015 May;24(5):349-53. doi: 10.1089/jwh.2015.5191. Epub 2015 Mar 31. PMID 25825986
- [Background] Quaife M, Cabrera M, Eakle R, Vickerman P, Delany-Moretlwe S, Terris-Prestholt F, editors. One size will not fit all: divergent stated preferences for new antiretroviral-based HIV prevention products across adults, adolescents and female sex workers in South Africa. EUHEA Conference: Hamburg, Germany; 2016.
- [Background] Quaife M, Eakle R, Cabrera Escobar MA, Vickerman P, Kilbourne-Brook M, Mvundura M, Delany-Moretlwe S, Terris-Prestholt F. Divergent Preferences for HIV Prevention: A Discrete Choice Experiment for Multipurpose HIV Prevention Products in South Africa. Med Decis Making. 2018 Jan;38(1):120-133. doi: 10.1177/0272989X17729376. Epub 2017 Sep 1. PMID 28863752
- [Background] Smith P, Tolla T, Marcus R, Bekker LG. Mobile sexual health services for adolescents: investigating the acceptability of youth-directed mobile clinic services in Cape Town, South Africa. BMC Health Serv Res. 2019 Aug 19;19(1):584. doi: 10.1186/s12913-019-4423-4. PMID 31426788
- [Background] Koss CA, Ayieko J, Mwangwa F, Owaraganise A, Kwarisiima D, Balzer LB, Plenty A, Sang N, Kabami J, Ruel TD, Black D, Camlin CS, Cohen CR, Bukusi EA, Clark TD, Charlebois ED, Petersen ML, Kamya MR, Havlir DV; SEARCH Collaboration. Early Adopters of Human Immunodeficiency Virus Preexposure Prophylaxis in a Population-based Combination Prevention Study in Rural Kenya and Uganda. Clin Infect Dis. 2018 Nov 28;67(12):1853-1860. doi: 10.1093/cid/ciy390. PMID 29741594
- [Background] Jamieson L, Johnson LF, Nichols BE, Delany-Moretlwe S, Hosseinipour MC, Russell C, Meyer-Rath G. Relative cost-effectiveness of long-acting injectable cabotegravir versus oral pre-exposure prophylaxis in South Africa based on the HPTN 083 and HPTN 084 trials: a modelled economic evaluation and threshold analysis. Lancet HIV. 2022 Dec;9(12):e857-e867. doi: 10.1016/S2352-3018(22)00251-X. Epub 2022 Nov 7. PMID 36356603
- [Background] Shah S, Hindley L, Hill A. Are New Antiretroviral Treatments Increasing the Risk of Weight Gain? Drugs. 2021 Feb;81(3):299-315. doi: 10.1007/s40265-020-01457-y. PMID 33400239